CLINICAL TRIAL: NCT01418885
Title: Correlation Exploration Between Cognitive Impairment and Neuroimaging and Inflammatory Markers in Patients With Subcortical Ischemic Vascular Disease
Brief Title: Cognitive Impairment , Neuroimaging and Inflammatory Markers in Patients With Subcortical Ischemic Vascular Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hebei General Hospital (Other)
Responsible Party: hebei general hospital, Neurology
Other Study IDs: dongyanhong85989995; Hebei general hospital (Other: Hebei general hospital)
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Other Generalized Ischemic Cerebrovascular Disease
Keywords: subcortical ischemic vascular disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- SIVD,VaD: vascular disease in patients with SIVD
- SIVD,VCIND: vascular cognitive impairment no dementia in patients with SIVD
- normal controls: normal elderly controls

SUMMARY:
SIVD is characterised by extensive cerebral white matter lesions (WML) and lacunar infarcts in deep grey and white matter structures. The relationship between SIVD and cognition is unclear, in part because of methodological inconsistencies across studies.

Diffusion tensor imaging (DTI) is a non-invasive water diffusion technique and can be used for quantitatively measuring the degree and directionality of the displacement distribution of water molecules. 1H magnetic resonance spectroscopy (1H-MRS) is a valuable tool for the assessment of several biochemical compounds in the brain in vivo, such as N-acetylaspartate (NAA), myoinositol (mI), Choline (Cho) and Creatine (Cr). There were few reports considering the relationship among MRS, DTI and cognitive impairment of SIVD. Combining MRS with DTI may provide valuable information about the pathophysiological changes underlying DTI abnormalities and help us to better understand the SIVD process. It has been proposed that the pathogenesis of SIVD related to cerebral small vessel disease caused by various mechanisms. Inflammation plays an important role in the pathogenesis of SIVD. The examination of inflammatory markers in relation to VaD might be benefit to early treatment.

In this study we applied neuropsychological tests, conventional MRI scanning, DTI, 1H-MRS techniques and inflammatory markers to estimate neuropsychological profile and white matter characteristics of imaging in patients with SIVD. Moreover, the relationship between WML and cognitive function impairment was also investigated. It could be possible to gain reliable data which is benefit to early diagnosis and treatment of cognitive impairment in SIVD.

DETAILED DESCRIPTION:
1. Contributions of white matter lesions to cognitive impairment in patients with subcortical ischemic vascular disease

   1. Extensive neuropsychological tests including MMSE and covering 5 cognitive domains including memory, executive, visuospatial, attention and language function would be performed on patients with SIVD and normal elderly controls matched in age and gender. The patients would be divided into VaD and VCIND group.
   2. Age-related white matter change rating scale, which is a visual rating scale developed by Wahlund, would be used to qualitative measure and locate the WML.
   3. Correlation analysis and hierarchical multiple regression analysis would be used to examine the relationship between general cognitive function and WML.
2. Evaluation of microstructural white matter lesions in patients with subcortical vascular cognitive impairment using diffusion tensor imaging

   1. SIVD patients divided into VaD and VCIND group and normal elderly controls matched in age and gender would be recruited. DTI images would be acquired, and fractional anisotropy (FA), mean diffusivity (MD) of normal-appearing white matter in cerebral lobes would be determined.
   2. These diffusion measurements were compared across the 3 groups, and significant differences would be further performed for correlation with tests of comprehensive cognitive function.
3. Evaluation of the lesions in thalamus and paraventricular white matter region in SIVD patients using 1H magnetic resonance spectroscopy and diffusion tensor imaging

   1. SIVD patients divided into VaD and VCIND group and normal elderly controls matched in age and gender would be recruited. The quantitative analysis of N-acetylaspartate (NAA), myoinositol (mI), Choline (Cho) and Creatine (Cr) resonance signals in region of interests located in thalamus and paraventricular white matter region would be measured. Ratios of NAA/ Cr, mI/ Cr and Cho/ Cr would be calculated in three groups.
   2. Conventional MRI and DTI scanning were received, FA and MD values of white matter in the same bilateral regions would be measured respectively.
   3. These diffusion measurements would be compared across the 3 groups, and significant differences would be further performed for correlation with tests of comprehensive cognitive function.
4. Clinical significance of serum inflammatory markers in SIVD patients

   1. SIVD patients divided into VaD and VCIND group and normal elderly controls matched in age and gender would be recruited. The serum levels of sCD40L, IL-6, hsCRP were detected by enzyme linked immunosorbent assay (ELISA) and fixed time nephelometry methods in all subjects, respectively.
   2. The relationship would be described among these inflammatory factors and WML, cognitive impairment in patients with SIVD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of subcortical ischemic vascular disease
* Must exist cognitive impairment

Exclusion Criteria:

* serious dementia could not speak , listen and white
* other diseases which might cause dementia

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with SIVD diagnosed according to the MRI criteria of Erkinjuntti ,25 normal elderly controls matched in age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Peiyuan Lv, Dr, Study Director — Hebei General Hospital
Locations (1):
- Yanhongdong, Shijiazhuang, Hebei, China

REFERENCES:
- See also: Links to Hebei general hospital web pages . — http://www.hbpphosp.cn